CLINICAL TRIAL: NCT01462032
Title: Training Executive, Attention, and Motor Skills (TEAMS): Preliminary Studies
Brief Title: Non-pharmacological Interventions for Preschoolers With Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: NIPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queens College, The City University of New York (Other)
Responsible Party: Principal Investigator, Jeffrey Halperin, Distinguished Professor of Psychology, Queens College, The City University of New York
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4R33MH085898-03 (NIH)
Record Dates: First submitted 2011-09-13; First posted 2011-10-28 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Preschool Children; ADHD; Treatment; Non-pharmacological
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive enhancing games (Experimental): Children will be introduced to specific games believed to enhance cognitive functioning. Parent will be encouraged to play these games with their children.
  Interventions: Behavioral: Training Executive, Attention and Motor Skills (TEAMS)
- Parent support and education (Active Comparator): Parents will participate in groups designed to provide information about ADHD and support for working with their child.
  Interventions: Behavioral: Parent support and education

INTERVENTIONS:
Behavioral: Training Executive, Attention and Motor Skills (TEAMS) — Children will be taught games targeting these skills and parents will be encouraged to play these games with children at home
  Arms: Cognitive enhancing games
Behavioral: Parent support and education — Parents will participate in groups designed to provide information about ADHD and support for working with their child.
  Arms: Parent support and education

SUMMARY:
This study is designed to evaluate two potential treatments for children with Attention-deficit/Hyperactivity Disorder (ADHD) that do not involve the use of medication. Our goal is to develop new interventions for preschoolers with ADHD that will result in enduring reductions of ADHD symptoms and associated impairments in children, and thus prevent long-term difficulties characteristic of many children with ADHD.

Both interventions involve weekly playgroups (of roughly five children) in which children engage in designated activities while parents engage in groups focusing on parent education, support, and their children's activities. It is hypothesized that both interventions will be helpful, but that only one will have lasting effects well beyond the end of active treatment.

DETAILED DESCRIPTION:
Children eligible for this study are:

* 4 and 5 years-old (between the ages of 48 - 72 months)
* shows signs and symptoms of hyperactivity, impulsiveness and/or inattention. To enter the study, following our evaluation, they will need to meet diagnostic criteria for ADHD
* enrolled in a preschool or daycare setting

Children are ineligible to participate in this study if they:

* are currently being treated with psychotropic medication
* have a diagnosed neurological disorder
* have an autism spectrum pr pervasive developmental disorder
* are intellectually impaired
* are highly physically aggressive

ELIGIBILITY:
Inclusion Criteria:

* Child is hyperactive
* Child meets criteria for ADHD
* Child attends preschool or kindergarten
* Family speaks English at home

Exclusion Criteria:

* Family does not speak English at home
* Child does not attend preschool/kindergarten
* Child is diagnosed with or suspected of having PDD
* Child has IQ of less than 80
* Child is being treated with psychotropic medication
* Child has a diagnosed neurological disorder
* Child is aggressive
* Child is only inattentive and does not exhibit signs of hyperactivity
* Parent has attended parent management classes
* Child is not physically able to participate in group play sessions

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2011-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Clinical Global Improvement Scale Rating at Post-Treatment, 1 Month, and 3 Months after Treatment | Assessed pre-treatment (@ 0 weeks), post-treatment (@ 5 weeks after treatment onset), 1-month follow-up (@ 9 weeks after treatment onset) and 3 months follow-up (@ 21 weeks after treatment onset)
  This is a clinical rating based on data derived from parent and teacher ratings as well as a semi-structured clinical interview with the child's caretaker.

SECONDARY OUTCOMES:
Change from Baseline Parent and Teacher Ratings on the ADHD-RS at Post-Treatment, 1 month, and 3 months after Treatment | Assessed pre-treatment (@ 0 weeks), post-treatment (@ 5 weeks after treatment onset), 1-month follow-up (@ 9 weeks after treatment onset) and 3 months follow-up (@ 21 weeks after treatment onset)
  These are parent and teacher ratings of ADHD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Halperin, Ph.D., Principal Investigator — Queens College, CUNY
Locations (1):
- Queens College, City University of New York, Flushing, New York, United States

REFERENCES:
- [Derived] Halperin JM, Marks DJ, Chacko A, Bedard AC, O'Neill S, Curchack-Lichtin J, Bourchtein E, Berwid OG. Training Executive, Attention, and Motor Skills (TEAMS): a Preliminary Randomized Clinical Trial of Preschool Youth with ADHD. J Abnorm Child Psychol. 2020 Mar;48(3):375-389. doi: 10.1007/s10802-019-00610-w. PMID 31834588